CLINICAL TRIAL: NCT04256304
Title: The Effect of The Personalized Patient Engagement Plan on Diabetes Management in Patients With Type 2 Diabetes
Brief Title: The Effect of The Personalized Patient Engagement Plan on Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Dilara Usta, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ka-19031
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Type 2 Diabetes; Patient Engagement; Self Efficacy; Adherence, Patient
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Participation; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Personalized Health Engagement Plan group
  1. First face-to-face session (Motivational interviewing) + Pre-tests
     * Patient Health Engagement Scale
     * Assessment Scale for Treatment Adherence in Type 2 Diabetes Mellitus
     * The Diabetes Management Self-Efficacy Scale for Patients with Type 2 Diabetes Mellitus
  2. Phone call coaching
  3. A set of personalized home-based exercises
  4. Second face-to-face session (Motivational interviewing) + Post-tests
  Interventions: Behavioral: PHEinAction-Personalized Patient Engagement Plan
- Control group (No Intervention): 1. First meeting (Pre-tests)
     * Patient Health Engagement Scale
     * Assessment Scale for Treatment Adherence in Type 2 Diabetes Mellitus
     * The Diabetes Management Self-Efficacy Scale for Patients with Type 2 Diabetes Mellitus
  2. Second meeting (Post-tests)
     * Patient Health Engagement Scale
     * Assessment Scale for Treatment Adherence in Type 2 Diabetes Mellitus
     * The Diabetes Management Self-Efficacy Scale for Patients with Type 2 Diabetes Mellitus

INTERVENTIONS:
Behavioral: PHEinAction-Personalized Patient Engagement Plan — The intervention includes two face-to-face sessions, a telephone consultation, and written home-based exercises. The first session aims to promote an awareness of patients with diabetes management, define an action plan to encourage engagement, introduce the patient to follow their strategy for the next four weeks, and encourage them to adopt the instruments with home-based exercises to reach their specified health goals. Two weeks after the first interview session, the researcher will provide telephone consultation to check the patient for their progress and support them to maintain motivation. The second session will include collecting patient's experiences and discussing the home-based exercises, re-determining the patient health engagement phase through the PHE-s®, discussing the personalized care goals by providing feedback aiming to support improvements, and setting a new engagement goal with the current status and encouraging the patient to maintain the health engagement plan.
  Arms: Intervention group

SUMMARY:
This study evaluates the effect of Personalized Patient Engagement Plan on diabetes management in patients with at least six months of Type-2 Diabetes. The research is planned to be carried out as an experimental study with pretest-posttest control groups.

Half of the participants will receive the Personalized Patient Engagement Plan; between two 2 face-to-face sessions including motivational interviews, one telephone coaching call and patient-driven home-based exercises will be conducted. Another half will receive usual care.

DETAILED DESCRIPTION:
Hypotheses

H1-1: Personalized Patient Engagement Plan will significantly affect the self-efficacy of patients with Type-2 Diabetes Mellitus.

H1-2: Personalized Patient Engagement Plan will significantly affect the treatment adherence of patients with Type-2 Diabetes Mellitus.

H1-3: Personalized Patient Engagement Plan will significantly affect the engagement levels of patients with Type-2 Diabetes Mellitus.

1. Patients who apply to the endocrine outpatient unit will be evaluated according to the inclusion and exclusion criteria. At first, the RA will obtain a daily list of patients waiting for their appointment with the endocrinologist each day of the recruitment period and will access the medical records of waiting patients and screen for the eligibility criteria. Patients meeting the eligibility criteria will be invited to a room located in the outpatient clinic and be asked to fill out Health Literacy Scale (HSL).
2. After the final eligibility assessment, the potential participants will be provided information regarding the study's objectives and be asked for their written informed consent. The researcher will collect consented participants' telephone numbers to determine their next endocrinologist appointment and collect the baseline data, including the sociodemographic and diabetes-related characteristics, laboratory HbA1c testing, body mass index (BMI), and the measures of treatment compliance, self-efficacy, and patient engagement.
3. Each participant will be assigned a number. In order to assign patients to the intervention and control groups, randomization will be carried out independently of the research via the link https://www.randomizer.org/.
4. After randomization is completed and participants are assigned to two groups, the application of the research will start. After this stage, defined interventions will be carried out for the intervention group. The Control group will only perform pre-post tests and receive usual care. The number of samples is expected to be 60, 30 for the intervention group and 30 for the control group. After these numbers are reached, a post power analysis will be done.

Independent variables; demographic characteristics of the patients (age, gender, marital status, employment status, educational status, presence of social security, economic status, place of residence, co-living, diabetes duration, type of treatment received, how long have been treated, experiencing chronic complications related to diabetes condition, acute complications due to diabetes, chronic disease other than diabetes, presence of diabetes disease in the family, monitoring status of blood sugar, regular exercise status, following diabetic diet status, if previously educated about diabetes disease, hospitalization due to diabetes condition, smoking status, alcohol use status, if receiving help to maintain diabetes treatment, and some parameters - body mass index, Hemoglobin A1c, total cholesterol, triglyceride, HDL, LDL, fasting blood sugar and satiety blood sugar) are independent variables.

Statistical analysis will be performed with SPSS 23 (IBM Inc, NY, USA). Correlation and regression will be applied for the mean scores of the scales, the differences between the two groups averages will be analyzed by the significance test of the difference between the two averages, the significance test of the difference between the two percentages, Mann-Whitney U or Chi-Square tests. The level of statistical significance of the study will be p <0.05. Depending on the normality of the data in dependent groups, a comparison will be made with the t-test or Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria:

* having type 2 diabetes for at least six months
* receiving medication for type 2 diabetes
* ability to speak, read, write and understand Turkish
* to score an average of 2.5 points on the Health Literacy Scale

Exclusion Criteria:

* being unable to take responsibility for self-care
* pregnancy/planning pregnancy
* severe thinking or mental problems (diagnosed psychiatric disorders).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Patient Health Engagement Scale | 1 month
  The Patient Health Engagement Scale (PHE-s) is an instrument assessing the engagement of patients in their care process and was developed in 2015 (Ordinal α=0,85). The PHE-s was developed based on the four-stage model of patient engagement (blackout, arousal, adhesion, and eudaimonic project), has an ordinal nature, and it consists of 5 items with seven responses, which allow patients' to reflect their experience about their care. In scoring, points 1 and 2 refer to the blackout, 3 and 4 to the arousal, 5 and 6 to the adhesion, and finally, point 7 refers to the eudaimonic phase. The median value is regarded while calculating the final PHE-s score. The Turkish validity study was conducted in 2019. The content validity index (CVI) was 0.98, and the Ordinal alpha was 0.80.
Assessment Scale for Treatment Adherence in Type 2 Diabetes Mellitus | 1 month
  The treatment adherence was assessed using the Assessment Scale for Treatment Adherence in Type 2 Diabetes Mellitus developed in 2017 for Turkish patients with diabetes, and Cronbach α was found to be 0,77. The scale consists of a total of 30 items and has a 5-point Likert structure (certainly agree=1, I agree=2, I partially agree=3, I do not agree=4, certainly do not agree=5). The highest score is 150 while the lowest score is 30. If the total score is between 30-54, it is considered as "good adherence"; if it is between 55-125, it is assessed "moderate adherence" and finally scores between 126-150 indicates "poor adherence" to the treatment. The scale consists of 7 sub-dimensions (emotional difficulties in compliance, physical difficulties in compliance, changing difficulties of habits in compliance, acceptance difficulties in compliance, awareness difficulties in compliance, diet difficulties in compliance, and denial difficulties in compliance).
The Diabetes Management Self-Efficacy Scale for Patients with Type 2 Diabetes Mellitus | 1 month
  The Self Effectiveness Scale for Diabetes Management in Type 2 Diabetes Patients was developed in 1999 to determine the level of self-efficacy they have during their care for diabetes patients.

OTHER OUTCOMES:
Health Literacy Scale for Turkish Diabetic Patients | 1 month
  Health Literacy Scale (HLS) for Turkish Diabetic Patients will be used for randomisation. The original HLS is comprised of three subscales to assess the functional (five items), interactive (five items), and critical (four items) health literacy of diabetes patients. The results of Turkish psychometric evaluation showed that the overall Cronbach's alpha for HLS was 0.96, and for functional, interactive and critical subscales were 0.96, 0.91, and 0.96, respectively, and S-CVI was 0.97. Higher scores in communicative and critical HL indicates higher HL, but the scores were reversed for the functional subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Fatoş Korkmaz, Assoc. Prof., Study Director — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University Faculty of Nursing, Ankara
  - Hacettepe University, Ankara

IPD SHARING:
Plan to Share IPD: Yes
IPD for all outcome measures will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Requestors will be required to sign a Data Access Agreement.